CLINICAL TRIAL: NCT01866631
Title: Using National University Cancer Institute of Singapore (NCIS) Registry to Measure Time Trends in Quality of Care for Breast Cancer Patients in a National Cancer Centre
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: BR08/30/10
Record Dates: First submitted 2012-10-31; First posted 2013-05-31 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
The investigators hypothesise that the research data will enable them to elucidate local clinical practices with regard to breast cancer care and enable them to extrpolate the data to improved local clinical care for their patients through self-regulation and audit.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 21 years old

Exclusion Criteria:

No patient involved

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To retropsectively review the NCIS registry of females diagnosed with breast cancer in years 2002 to 2008 with regards to clinical quality indicators as published by the European Sociaty of Breast Cancer Oncologists (Eur J Can 2010; 46:2344-2356). We will extract data from a pre-existing breast cancer registry which belongs to NCIS, looking at data which includes the following:(1) Completeness of clinical and imaging diagnostic work-up(2) Completeness of prognostic and predictive characterization(3) Multidisciplinary discussion(4) Appropriate surgical approach(5) Appropriate post-operative radiation(6) Avoidance of over-treatment(7) Appropraiet hormonal therapy(8) Appropriate chemotherapy and other medical therapy(9) Staging, counselling, follow-up and rehabilitative procedures
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Quality of care at NCIS using indicators | 2 years

SECONDARY OUTCOMES:
The trends and variations in quality of care indices over a period of years | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore